CLINICAL TRIAL: NCT06846242
Title: Validity and Reliability of the Scapular Muscular Endurance Test in Adolescents
Brief Title: Validity and Reliability of the Scapular Muscular Endurance Test
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Lecturer, Istinye University
Other Study IDs: 24-30
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Scapular Muscle Endurance; Adolescent
Keywords: Assessment; Performance; Upper Extremity; Psychometric Properties
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Adolescents
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The group in which the assessments will be made.

SUMMARY:
The scapula plays a crucial role in proper shoulder function, contributing to synchronized scapular rotation during humeral motion, serving as a stable base for rotator cuff activation, and acting as a key link in the kinetic chain. Each of these functions is essential for optimal arm movement and depends on the integrity of the surrounding shoulder anatomy. However, bone and soft tissue damage, as well as muscle weakness and shortening, can alter the scapula's roles, affecting both its resting position and dynamic motion. This altered scapular position and/or motion is referred to as scapular dyskinesia.

Although scapular dyskinesia is commonly observed in shoulder injuries, it is generally considered a nonspecific response to shoulder pain rather than a direct consequence of a specific glenohumeral pathology. Therefore, assessing the presence or absence of scapular dyskinesia is a critical component of clinical evaluation. A comprehensive assessment should include a visual examination of the scapula at rest and during dynamic humeral movements, as well as objective measurements of posture and the performance of scapular corrective maneuvers. These evaluations assist clinicians in determining the extent to which scapular involvement contributes to a given shoulder injury.

The treatment of scapular dyskinesia should begin with optimizing anatomical alignment, followed by restoring dynamic scapular stability through the strengthening of scapular stabilizers using kinetic chain-based rehabilitation protocols. The kinetic chain, as defined by Steindler, is "a combination of successive joints containing complex motor units." It describes the interconnected movement of joints, where adjacent segments interact to form a continuous chain of motion. This biomechanical model emphasizes that dysfunction in any part of the chain can impact movement quality in both upper and lower segments. The scapula is a foundational component within this system, with surrounding muscles playing a crucial role in stabilizing it.

Postural disorders such as kyphosis can lead to scapular deformities, negatively affecting scapular stability. Rehabilitation professionals and researchers increasingly use the Scapular Muscular Endurance Test (SMET) to assess scapular stability. Given that adolescents are at a heightened risk for musculoskeletal injuries, upper extremity assessments like the SKET may contribute significantly to evaluating this population. However, the validity and reliability of the SMET in adolescents have yet to be established.

This study aims to determine the validity and reliability of the SKET in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Being between 10-19 years old
* Being willing to participate in the study

Exclusion Criteria:

* Those who have had major surgery or trauma related to the musculoskeletal system, especially the upper extremity and scapular region
* Those with neurological diseases
* Those with rheumatic diseases in the active phase
* Those with systemic diseases (Diabetes, hypothyroidism, infection, malignancy...)

Ages: 10 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents between the ages of 10-19 will be included.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Scapular Endurance Test | 2 weeks
  The endurance of the scapular muscles will be evaluated with the Scapular Muscular Endurance Test (SMET). The SMET will be performed with the participants standing facing the wall, with the shoulders and elbows in a 90° flexion position. When both scapulae are in a neutral position, the most suitable length of 10 wooden bars of different lengths (18-36 cm) will be placed between the participant's elbows and a dynamometer will be placed between the participant's hands. In this position, the participant will be asked to perform shoulder external rotation until a load of one kilogram is reached on the dynamometer and to maintain this force, and the results will be recorded in seconds. The time the participant meets the test conditions will be recorded in seconds with a stopwatch. The test will be repeated twice with a five-minute break for rest, with the best score recorded for analysis.
Closed Kinetic Chain Upper Extremity Stability Test | 2 weeks
  It will be used to evaluate upper extremity strength, endurance, and closed kinetic chain. The test will be performed following the instructions defined by de Oliveira et al. During the test, male participants will be placed in a push-up position and female participants in a modified push-up position (with knee support) on 2 tapes attached to the floor with a distance of 90 cm between their hands. Participants will be asked to touch their other hand with one hand while maintaining the push-up position for 15 seconds and the number of repetitions completed for the right and left will be recorded. The test will be repeated three times and the average of the values will be recorded. 45-second rest breaks will be given between each test.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided